CLINICAL TRIAL: NCT04716322
Title: Study of the Determinants Associated With Sustained Changes in Physical Activity Behaviors, and Their Effects on the Prevention and Treatment of Chronic Diseases, in Individuals Enrolled in an Adapted Physical Activity Program
Brief Title: Health-Enhancing Adapted Physical Activity Program at "Mon Stade"
Acronym: SESAME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mon Stade Sports Medicine Centre (Other)
Collaborators: Laboratory MOVE, Faculty of Sport Sciences, University of Poitiers, France (Unknown); Public Health Foundation of MGEN, France (Unknown); General Mutual Insurance of National Education, France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-A00254-35
Record Dates: First submitted 2020-12-23; First posted 2021-01-20 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Exercise Therapy; Behavior and Behavior Mechanisms; Adherence, Patient; Lifestyle, Sedentary; Life Style; Life Style, Healthy; Cost-Benefit Analysis; Prescriptions; Physical Activity; Adapted Physical Activity
Keywords: Adapted Physical Activity; Active Live Habits; Adherence; Aerobic Capacity; Behavior; Body Composition; Budget Impact Analysis; Cardiorespiratory Fitness; Care Consumption; Chronic Disease; DEXA scan; Exercise; Health-Adapted Physical Activity; Health-Enhancing; Life-Style; Long-Term Illness; Medico-Economic; Motivation; Perceived Barriers; Physical Activity; Physical Fitness; Prescription; Prevention; Psycho-social; Quality Of Life; Questionnaire; VO 2 measurement
MeSH Terms: conditions — Behavior; Patient Compliance; Sedentary Behavior; Motor Activity; Chronic Disease

STUDY DESIGN:
Intervention Model Description: Prospective monocentric cohort with consecutive inclusions of participants with chronic disease, and followed for 5 years after an initial 16-week physical activity program intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted Physical Activity (Other): A 16-week health-adapted physical activity program and 5-year follow-up
  Interventions: Behavioral: Adapted Physical Activity

INTERVENTIONS:
Behavioral: Adapted Physical Activity — A 16-week health-adapted physical activity program, individualized from baseline evaluation of participants including the specificities of their pathologies

SUMMARY:
Introduction: Regular practice of exercise or physical activity (PA) is a recognized intervention as a determinant of good health acquisition, maintenance, or recovery for a large number of chronic pathologies. Nevertheless, few studies have evaluated adherence to an initial health-adapted PA (APA) program, and persistence of active behavior over the time in individuals with a chronic disease.

The aim of the study is to determine the brakes and levers associated with motivation and long-term compliance. In addition, the investigators aim to evaluate the cost-effectiveness of such program in term of care consumption. Finally, the investigators complete their interest for APA prescription from practitioners agreeing to enroll their patients in the present study.

Method: The investigators perform a prospective monocentric cohort, of 2024 patients affected of a chronic disease or long-term illness (LTI), enrolled from 2021 to 2024 (4 years, 506 per year), for a 16-week APA program, and followed 5 years with an annual fitness and habits of life and care consumption evaluation.

DETAILED DESCRIPTION:
Background:

While physical inactivity is the first modifiable risk factor (2nd is tobacco consumption) for cardiovascular morbidity and mortality and cancer in the World, regular physical activity (PA) is a recognized intervention with a high level of evidence, as a key determinant of good health acquisition, maintenance, or recovery for a large number of chronic pathologies.

The following 3 points caught the investigators' interest:

Point n°1: The 2019 collective expertise of the French National Institute of Health and Medical Research (INSERM) "Physical Activity: Prevention and Treatment of Chronic Diseases" reported following findings on the motivational aspects of regular or non-regular PA practice by people suffering from a chronic disease: 1) people with chronic disease practice less than the general population of the same age; 2) a significant number of patients do not participate in the proposed PA programs, and high drop-out rates are reported during these programs; 3) only a small percentage of patients maintain PA after completion of these programs. However, there is a lack of evidence and inconsistent quality studies regarding changes in duration of behavior following PA intervention programs. Follow-up of behavioral changes beyond 2 years is extremely rare in the literature. Thus, the problem is of a behavioral nature: on one hand, whether or not a person with a chronic disease adheres to an initial health-adapted PA program (APA), and on the other hand, whether or not a PA practice persists or is maintained over time. The identification of barriers and levers is key to help define actionable means to support adherence and enhance the sustainability of the virtuous behavior change induced by an initial program. This need for studies is underlined by "The group of experts [from INSERM, which] recommends: 1) long-term intervention studies with supervised exercises and 2) long-term post-intervention follow-up in order to better evaluate the continuation of program practice in autonomy", but also "to promote research on motivation and long-term compliance".

Point n°2: In relation to the benefit of PA programs on the physical and psycho-social fitness of individuals, the effects on health are demonstrated. As a result, a decrease in the prevalence of health events and their complications can be observed, as well as a more detailed use of care (drug treatment, consultations, and hospitalizations) depending on whether or not the participant benefits from an APA intervention. The medico-economic impact of such APA intervention has been little studied. Thus, the problem is of a medico-economic nature: the interest will initially focus on the evolution of care pathways over time, and the differences observed according to pathologies, but also according to the participants' behavior, in terms of compliance, or persistence or not in the duration of the favorable change in behavior initially acquired. An evaluation of care consumption and care pathways according to whether individuals have benefited from an APA program as proposed (SESAME cohort) or not (controls) also appears justified and will come later. This need for studies is emphasized by the INSERM expert group, which recommends "evaluating the cost-effectiveness of interventions according to the technique(s) used".

Point n°3: While the attending physician can prescribe an APA program to his patients with a chronic disease through a list of 30 long-term illness (LTI), (Article L. 1172-1 of the French Public Health Code and Decree N° 2016-1990 of December 30, 2016), the practitioner is confronted on the one hand with chronic pathologies outside of LTI list for which APA provides a demonstrated benefit (arterial hypertension (HTN), obesity, chronic obstructive pulmonary disease (COPD)), and on the other hand with a lack of experience in this non-medicinal prescription. Thus, the problem is of an operational practical nature in the prescription of APA, with a need for collection and analysis of the brakes and levers that can be applied to the prescription of APA, and for training and coordination of medical actors with APA professional. This need is underlined by the INSERM expert group, which recommends "the development of exchanges and joint reflection between the different professions involved in favor of the practice of APA."

Objectives:

In view of all these elements, the SESAME project consists in the prospective constitution of a cohort of people affected by a chronic pathology and enrolled in a 16-week individualized, educational and structured APA program, with a 5-year follow-up, providing support for an observational study whose main objective is the behavioral analysis of the brakes and levers associated with the persistence over time of a favorable change in behavior induced by an initial APA program.

Secondary objectives are: 1) an analysis of the effects of the program on the physical and psychological fitness parameters; 2) a behavioral analysis of the brakes and levers associated with good adherence to the initial APA program; 3) a medico-economic analysis: a) volume-based care consumption analysis: monitoring the evolution of the participants' care pathway and care consumption over time; b) cost analysis: expressing care consumption in monetary units; c) budget impact analysis: estimating the difference in costs between the "APA strategy" for SESAME participants and the "usual care strategy" of members of the French health insurance "Mutuelle Générale de l'Education Nationale" (MGEN) with comparable characteristics in terms of age and gender and belonging to the following subgroups; 4) an analysis of the practice of prescribing APA among physicians, and their brakes and levers for such a prescription.

Methods:

Prospective and consecutive constitution of a monocentric cohort, for the behavioral and medico-economic analysis of the effects of a non-medicinal intervention by the APA (qualified as a research involving the human person type 2 "RIPH 2" within the meaning of article L. 1121-1 of the French Public Health Code).

Duration of the inclusion period: 4 years Duration of follow-up for the participant: 5 years Number of visits for participant: 7 (Inclusion; end of 48 sessions of APA program over 16 weeks (maximum 9 months from start); at 1 year; 2 years; 3 years; 4 years and 5 years) Number of participants: 2024 (506 per year) Due to the lack of behavioral studies in population of individuals with a chronic condition for which the benefit of APA has been demonstrated, the number of subjects required cannot be calculated. Given the experience of a 1st pilot cohort of 600 people with chronic pathologies (including obesity) treated with support from the Regional Health Agency (ARS) Île-de-France in 2014-2016, a number of 2024 people for the constitution of the SESAME cohort is feasible, with a recruitment of 506 participants per year for 4 years.

The participants will be recruited consecutively according to the terms of the French Law (Decree n°2016-19990 of 30 Dec 2016, entered into application on 01 March 2017) relating to the conditions of dispensation of APA prescribed by the attending physician to patients suffering from LTI. For the study, the pathology criteria are extended to chronic pathologies outside 30-LTI list for which the benefit of APA has been demonstrated with a high level of evidence (grade A) including, among others, obesity, HTN, COPD, as well as to the sequelae of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection in the context of coronavirus 2019 disease (COVID-19). According to the prescription of his doctor, the patient will go to "Mon Stade" Sport Medicine Center, and will benefit from inclusion in the program.

The measurements, collections, health examinations and follow-up of the participants will be carried out by the personnel of "Mon Stade" (doctors and physical preparers/teachers in APA, APA master trainees and doctoral students, administrative or paramedical agents) according to their fields of competence and prerogatives. They will receive a specific training on how to pass questionnaires and tests in order to standardize data collection and to know the course of care for these evaluations.

The APA program has been established according to a standardized, homogenous, shared and coordinated practice protocol by all the operators, for each stage of the course: inclusion of the participant, initial evaluation, design, supervision and monitoring of the training plan, and final evaluation. The 16-week program consists of 3 sessions per week, including 2 supervised sessions with individualized educational follow-up by a physical trainer (MSc Sport Sciences, specialized in APA) at "Mon Stade", and 1 session in autonomy (can be done at home). Each session includes: a warm-up phase with articular and muscular awakening carried out autonomously; a 1-hour session bodywork combining 25 minutes of interval aerobic exercises (split type) and 25 minutes of neuromuscular reinforcement in circuit. The intensities and modalities of the exercises will have been personalized according to the results of the initial fitness assessment.

Regarding the behavioral analysis, the characteristics of physical and mental condition, quality of life and behavior will be observed as a function of time, and compared according to the following subgroups: 1) General characteristics: gender, age group, body mass index (BMI), socioeconomic category, childhood lifestyle habits, history of participation in an APA program; 2) Chronic disease groups for inclusion: metabolic (obesity, diabetes); cardiovascular-renal (HTN, coronary artery disease, heart failure, arteritis, stroke, kidney disease); respiratory (COPD, asthma, cystic fibrosis); oncological (solid and non-solid neoplasia); neurological (epilepsy, Parkinson's, Alzheimer's); psychiatric (depressive syndrome, bipolarity, schizophrenia); osteoarticular (chronic low back pain, chronic inflammatory rheumatism, arthritis, osteoporosis); infectious (human immunodeficiency virus (HIV), viral hepatitis C, SARS-CoV-2); 3) Observer" vs. "non-observer" status in the initial APA program, with collection of data on program attendance, the number of sessions carried out in a supervised manner at "Mon Stade" or independently (declarative), the actual duration of the program, and the reasons for its possible interruption ("Observers" = ≥90% completion of the 2 weekly supervised sessions of the initial APA program over a period of 4 to 9 months); 4) "Persistent" vs. "Non-persistent" status at 1, 2, 3, 4 and 5 years regarding the favorable behavior change initially acquired ("Persistent" = participants with a positive trajectory of the percentages of "moderate to vigorous" PA collected each year by wearing an accelerometer over 7 days).

Medico-economic analysis includes: 1) an analysis of care consumption by volume (consumption and care pathway over time); comparison by subgroups of participants; 2) a cost analysis; average cost by subgroups of participants compared to overall cost; 3) a budget impact analysis by estimating the difference in costs between SESAME participants and MGEN members with comparable age and gender characteristics who follow the usual care strategy among LTI, hypertensive, and obese patients.

Analysis of APA prescribing practice includes: 1) a phase of identification of potential prescribing practitioners from Parisian centers likely to refer patients; 2) an analysis of the general characteristics of practitioners, as well as their PA level by questionnaire; 3) an analysis of their barriers and levers to the practice of PA; 4) an analysis of their barriers and levers to the prescription of APA with a questionnaire dedicated to this objective; 5) the participatory development of the prescription and patient follow-up tools.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years of age or older
* Speaking and understanding French
* Affected by a chronic pathology according to a predefined list (LTI, obesity, HTA, COPD, COVID-19 with persistent symptoms)
* Carrier of a writing APA prescription
* Able to come to "Mon Stade" twice a week for their APA sessions following the 16-week health-adapted PA program;
* Signature of the information and consent form.

Exclusion Criteria:

- Women whose pregnancy is known

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2024 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year persistence of a positive trajectory of active behavior | 5 years
  Study of the brakes and levers associated with the persistence at 5 years of an initial 16-week APA program, of a positive trajectory of the percentages of "moderate to vigorous" AP practice collected by wearing for 7 days a wGT3X-BT type accelerometer (Actigraph, Pensacola, FL, USA), illustrating the persistence of the favorable change in behavior eventually induced

SECONDARY OUTCOMES:
Behavioral analysis: Lifestyle habits: Accelerometer: Daily sedentary time | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Changes in daily sedentary time (min) measured by wearing on the belt over 7 days an accelerometer "Actigraph wGT3X-BT"
Behavioral analysis: Lifestyle habits: Accelerometer: Time in sitting, standing or lying down | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Changes in Time in sitting, standing or lying down (min) measured by wearing on the belt over 7 days an accelerometer "Actigraph wGT3X-BT"
Behavioral analysis: Lifestyle habits: Accelerometer: Number of steps | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Changes in number of steps (n) measured by wearing on the belt over 7 days an accelerometer "Actigraph wGT3X-BT"
Behavioral analysis: Lifestyle habits: Accelerometer: Average daily energy expenditure (KCal) | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Changes in average daily energy expenditure (MET-min per day) measured by wearing on the belt over 7 days an accelerometer "Actigraph wGT3X-BT"
Behavioral analysis: Lifestyle habits: Global Physical Activity Questionnaire "GPAQ" | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Changes in average daily energy expenditure (MET-min per day) assessed by the Global Physical Activity Questionnaire "GPAQ" version 2
Behavioral analysis: Lifestyle habits: "Ricci & Gagnon" | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Changes in average score of "Ricci & Gagnon" physical activity questionnaire (6-9: Not active; 10-18: Weakly active; 19-27: Moderately active; 28-36: Active; 37-45: Very active)
Behavioral analysis: Lifestyle habits: "Ricci & Gagnon" vs. GPAQ | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Corelation between average score of "Ricci & Gagnon" questionnaire and average daily energy expenditure (MET-min per day) assessed by the Global Physical Activity Questionnaire "GPAQ" version 2
Behavioral analysis: Lifestyle habits: "Ricci & Gagnon" vs. Accelerometer | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Corelation between average score of "Ricci & Gagnon" questionnaire and average daily energy expenditure (MET-min per day) measured by wearing on the belt over 7 days an accelerometer "Actigraph wGT3X-BT"Activity Questionnaire "GPAQ" version 2
Behavioral analysis: Quality of life, psychological determinants: Eating habits | End of the APA program (between 4 and 9 months), 5 years
  Changes in quality of eating habits using a dedicated questionnaire
Behavioral analysis: Quality of life, psychological determinants: Alcohol consumption | End of the APA program (between 4 and 9 months), 5 years
  Changes in quantity consumption of alcoholic beverages using a dedicated questionnaire
Behavioral analysis: Quality of life, psychological determinants: Sleep | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Changes in quality of sleep using a dedicated questionnaire
Behavioral analysis: Quality of life, psychological determinants: WHOQOL-BREF | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Changes in 4-class scores of World Health Organisation Quality of Life "WHOQOL-BREF" questionnaire (1. Physical Health; 2. Psychological Health; 3. Social Relations; 4. Environment)
Behavioral analysis: Quality of life, psychological determinants: POMS | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Changes in 7-class T-scores of Profile of mood states "POMS" questionnaire (1. anxiety; 2. anger; 3. fatigue; 4. Vigor; 5. Depression; 6. Confusion; 7. Interpersonal relationship)
Behavioral analysis: Quality of life, psychological determinants: EMAPS | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Changes in 6-class scores of Health Purpose Physical Activity Motivation Scale "Echelle de Motivation envers l'Activité Physique en contexte de Santé" "EMAPS" including the six forms of motivation underlined by self-determination theory (1. Intrinsic motivation; 2. Extrinsic motivation - integrated; 3. Extrinsic motivation - identified; 4. Extrinsic motivation - introjected; 5. Extrinsic motivation - external regulation; 6. Amotivation)
Behavioral analysis: Quality of life, psychological determinants: QBAP | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Changes in 7-class scores of Barriers to Physical Activity Practice Questionnaire "Questionnaire des Barrières à la Pratique d'ACtivité Physique" "QBAP" (1. Personal operation; 2. Social Support; 3. Temporal organization; 4. Knowledge and information; 5. Accessibility; 6. Skills, personality; 7. Disinterest)
Behavioral analysis: Parameters associated with good adherence to the initial APA program | End of the APA program (between 4 and 9 months)
  Good adherence defined by a ≥90% completion of the 2 weekly supervised sessions of the initial APA program over a period of 4 to 9 months
Behavioral analysis: Parameters associated with persistence of physical activity practice over time | 1 year, 2 years, 3 years, 4 years
  Persistence of physical activity (PA) practice defined by the observation of a positive trajectory of "moderate to vigorous" PA practice percentages collected by wearing an accelerometer for 7 days
Medico-Economic Analysis: Care consumption | 1 year, 2 years, 3 years, 4 years, 5 years
  Changes in the volume of care consumption by subgroups of diseases using a dedicated questionnaire
Medico-Economic Analysis: Cost of the APA program: Direct costs | 1 year, 2 years, 3 years, 4 years, 5 years
  Cost of the program and care consumption (hospitalizations, consultations, medications) using a dedicated questionnaire
Medico-Economic Analysis: Cost of the APA program: Indirect costs | 1 year, 2 years, 3 years, 4 years, 5 years
  Monetary evaluation of caregivers' time for informal care, absenteeism, opportunity cost of the program for patients, using a dedicated questionnaire
Medico-Economic Analysis: Budget impact analysis | 1 year, 2 years, 3 years, 4 years, 5 years
  Budget impact analysis (BIA) of the APA program, which will mobilize MGEN medical-administrative and survey data, in order to estimate the difference in cost between SESAME cohorts and MGEN members who do not benefit from an APA, for population subgroups that are comparable in terms of age group and gender and according to their chronic diseases
Analysis of APA prescription: | During the 4 years of participants' inclusion for the study
  Analysis of APA prescription using a dedicated questionnaire of perceived barriers to the medical prescription of APA

OTHER OUTCOMES:
Effects on physical fitness: General measures: Weight | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Body mass (Kg) measured on a balance
Effects on physical fitness: General measures: Body mass index "BMI" | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  BMI (Kg/m²) = Weiht/(Height)²
Effects on physical fitness: General measures: Waist circumference | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Waist circumference (cm) measured in standing position with a tape measure
Effects on physical fitness: General measures: Resting blood pressure | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Blood pressure (BP) measured after 5 minutes rest in lying position (mm Hg) with an automatic BP device
Effects on physical fitness: General measures: Resting heart rate | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Heart rate after measured after 5 minutes rest in lying position (mm Hg) with the automatic BP device
Body composition: DEXA scan: Fat mass | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Total fat mass (g) measured with the DEXA scan
Body composition: DEXA scan: Visceral fat mass | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Visceral fat mass (cm²) measured with the DEXA scan
Body composition: DEXA scan: Lean mass | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Total lean mass (g) measured with the DEXA scan
Body composition: DEXA scan: Bone mass | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Total bone mass (g) measured with the DEXA scan
Body composition: Impedance meter: Intracellular water | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Volume of total body intracellular water (L) measured with the impedance meter
Body composition: Impedance meter: Extracellular water | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Volume of total body extracellular water (L) measured with the impedance meter
Respiratory capacity (spirometry): Forced vital capacity "FVC" | 5 years
  Forced vital capacity (L) measured by spirometry before the cardiorespiratory exercise test
Respiratory capacity (spirometry): Forced expiratory volume in 1 second "FEV1" | 5 years
  Forced expiratory volume in 1 second (L) measured by spirometry before the cardiorespiratory exercise test
Respiratory capacity (spirometry): Peak expiratory flow "PEF" | 5 years
  Peak expiratory flow (L/min) measured by spirometry before the cardiorespiratory exercise test
Aerobic capacity (exercise stress test): Maximum aerobic power "MAP" if performed on Ergo-cycle | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Maximum aerobic power (Watts) measured by a maximum incremental stress test performed on an ergo-cycle
Aerobic capacity (exercise stress test): Maximum aerobic speed "MAS" if performed on Treadmill | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Maximum aerobic speed (km/h) measured by a maximum incremental stress test performed on a treadmill
Aerobic capacity (exercise stress test): METs max | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  METs max (METs) estimated by a maximum incremental stress test performed either on an ergo-cycle nor on a treadmill
Aerobic capacity (exercise stress test): Heart rate max | End of the APA program (between 4 and 9 months), 1 year, 2 years, 3 years, 4 years, 5 years
  Heart rate max (beats/min) measured by a maximum incremental stress test performed either on an ergo-cycle nor on a treadmill
Aerobic capacity (exercise stress test): V'O2 max | End of the APA program (between 4 and 9 months), 5 years
  V'O2 max (L/min) measured by a maximum incremental cardiorespiratory stress test performed either on an ergo-cycle nor on a treadmill
Neuromuscular capacity: Maximum strength of lower limbs | End of the APA program (between 4 and 9 months), 5 years
  Maximum strength of lower limbs (Kg) measured on a leg-press "Keiser® Air 420"
Neuromuscular capacity: Maximum strength of upper limbs | End of the APA program (between 4 and 9 months), 5 years
  Maximum strength of upper limbs (Kg) measured on a leg-press "Keiser® Air 420"
Neuromuscular capacity: Lumbar muscular endurance | End of the APA program (between 4 and 9 months), 5 years
  Lumbar muscular endurance using Sorensen Test (sec)
Neuromuscular capacity: Abdominal muscular endurance | End of the APA program (between 4 and 9 months), 5 years
  Abdominal muscular endurance using Shirado-Ito Test (sec)
Neuromuscular capacity: Handgrip | End of the APA program (between 4 and 9 months), 5 years
  Static handgrip strength test with a dynamometer (Newton)
Neuromuscular capacity: Balance | End of the APA program (between 4 and 9 months), 5 years
  One leg balance using Flamingo Balance Test (sec)
Neuromuscular capacity: Flexibility | End of the APA program (between 4 and 9 months), 5 years
  Trunk flexibility test using Sit-And-Reach Test (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Sosner, MD, PhD, Study Director — Mon Stade Sports Medicine Center, Paris, France
Locations (1):
- Mon Stade Sports Medicine Center, Paris, France

IPD SHARING:
Plan to Share IPD: No